CLINICAL TRIAL: NCT03715842
Title: Clinical Assessment Of Inlay Retained Bridge Designs (Tub Shaped And Inlay Shaped) In Missing Posterior Teeth Cases.
Acronym: dentistry
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, mahmoud osama, clinical professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEBD-CU-2018-10-08
Record Dates: First submitted 2018-10-10; First posted 2018-10-23 (Actual); Last update posted 2018-10-23 (Actual); Status verified 2018-10

CONDITIONS: Missing Tooth
MeSH Terms: conditions — Anodontia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tub shaped design (Experimental): The tub-shaped preparation design this consists of an occlusal proximal reduction featuring a 3.5-4 mm width bucco-lingually, 3-3.5mm depth occluso-gingivally and 7-7.5 mm length mesio distally for molars and 2.3-2.8mm width buccolingually, 3-3.5 mm depth occluso gingivally and 3.5-4mm length mesiodistally for premolars. when necessary, superficial extensions may also be made on the preparations so that the occlusal fossa included in the preparation area and then the susceptibility for plaque accumulation will be diminished.
  Interventions: Other: Tub shaped design
- Inlay shaped design (Active Comparator): The occlusal inlay had a preparation depth that allowed a thickness of 2.0 mm for the ceramic. The occlusal preparation was 4 mm wide and extended 4 or 6 mm mesio-distally for the premolar or molar models, respectively. The proximal box was 1 mm wide and had approximately 5˚ divergence, extending 2 mm apical to the isthmus floor . The preparations corresponded to a proximal connector area of 3 mm × 3 mm for molars and premolars.
  Interventions: Other: Inlay shaped design

INTERVENTIONS:
Other: Tub shaped design — The tub-shaped inlay preparation design this consists of an occlusal proximal reduction featuring a 3.5-4 mm width bucco-lingually, 3-3.5mm depth occluso-gingivally and 7-7.5 mm length mesio distally for molars and 2.3-2.8mm width buccolingually, 3-3.5 mm depth occluso gingivally and 3.5-4mm length mesiodistally for premolars. when necessary, superficial extensions may also be made on the preparations so that the occlusal fossa included in the preparation area and then the susceptibility for plaque accumulation will be diminished.
  Arms: Tub shaped design
Other: Inlay shaped design — The occlusal inlay had a preparation depth that allowed a thickness of 2.0 mm for the ceramic. The occlusal preparation was 4 mm wide and extended 4 or 6 mm mesio-distally for the premolar or molar models, respectively. The proximal box was 1 mm wide and had approximately 5˚ divergence, extending 2 mm apical to the isthmus floor . The preparations corresponded to a proximal connector area of 3 mm × 3 mm for molars and premolars.
  Arms: Inlay shaped design

SUMMARY:
The interest in partial coverage retainers such as inlays and onlays have increased drastically because these restorations are able to provide a more conservative option requiring minimal tissue removal thus preserving healthy tooth structure to a maximum extent.

If patient rejects an implant treatment and enough sound tooth structure is available it would be desirable to restore a missing tooth with Inlay-Retained Fixed Partial Denture instead of full coverage retained one .

The use of all-ceramic materials for inlays and onlays in restorative dentistry is becoming more popular , the proper selection of restorative materials, careful preparation design and adequate adhesion between tooth/restorative material interfaces considered important factor to prevent failures .

Zirconia was introduced into dentistry in the 1990s.The high initial strength and fracture toughness of zirconia results from a physical property of partially stabilized zirconia known as transformation toughening. On the other hand, its white color, similar to the color of natural teeth and its ability to transmit light makes it useful in aesthetically important areas .

Inlay Fixed Partial Denture restoration may have increased the risk of fracture due to the relative small size of restorations compared to the complete coverage restoration. An unfavorable distribution of stresses between the ceramic inlay and tooth structure may result in marginal deterioration around the inlay or its failure.

The direction of forces on the occlusal surface of Inlay Fixed Partial Denture may lead to the phenomenon of submargination, ceramic fracture, wear at interface and postoperative hypersensitivity which remain a problem that require further investigation. One of the most important factors in the success and longevity of a restoration is to have an accurate marginal fit. Ideally, the cemented restoration should precisely meet the finish line of the prepared tooth. In reality, clinical perfection is challenging to achieve and to verify.

DETAILED DESCRIPTION:
The tub-shaped inlay preparation design this consists of an occlusal proximal reduction featuring a 3.5-4 mm width bucco-lingually, 3-3.5mm depth occluso-gingivally and 7-7.5 mm length mesio distally for molars and 2.3-2.8mm width buccolingually, 3-3.5 mm depth occluso gingivally and 3.5-4mm length mesiodistally for premolars. when necessary, superficial extensions may also be made on the preparations so that the occlusal fossa included in the preparation area and then the susceptibility for plaque accumulation will be diminished.

Participant timeline

The visits will be designated as follows:

Visit 1: one week after allocation, preoperative records, face-to-face adherence reminder session, clinical examination, radiographic examination, intraoral photography and primary impressions for diagnostic cast construction .

Visit 2: one week after the first visit, teeth preparations, secondary impression and temporization .

Visit 3: one week after the second visit, try in for the restoration will be done.

Visit 4: one week after the try in, final cementation of the restoration.(GC resin cement) Visit 5: follow up after twelve months from the cementation visit.

The aim of the study is to assess the fracture resistance of two inlay retained bridge designs (tub shaped and inlay shaped) in missing posterior teeth cases. Based on previous papers by Ohlmann et al., 2008 7 and İzgi et al.,2011 4 indicate that the failure rate among controls is 52%. If the true failure rate for experimental subjects is 99%, we will need to study 12 in each group to be able to reject the null hypothesis that the failure rates for experimental and control subjects are equal with probability (power) 0.8. The Type I error probability associated with this test of this null hypothesis is 0.05. We will use an uncorrected chi-squared statistic to evaluate this null hypothesis. This number is to be increased to 15 in each group (25% more than the calculated) to compensate for possible losses during follow up. The sample size was calculated by PS: Power and Sample Size Calculation software Version 3.1.2 (Vanderbilt University, Nashville, Tennessee, USA).

ELIGIBILITY:
Inclusion Criteria:

* From 18-55 years old, should be able to read and sign the consent document.
* Ability to tolerate the restorative procedures (physical and psychological).
* Good oral hygiene
* Low susceptibility to decay
* Have a minimum coronal tooth height of 5 mm,
* Parallel abutments
* Sufficient mesio distal edentulous gap dimensions.

Exclusion Criteria:

* Partially erupted teeth (young)
* Bad oral hygiene and motivation
* Root canal treated teeth
* Psychiatric problems or unrealistic expectations
* Severe para-functional habits
* The absence of enamel on the preparation margins
* Extensive crown defects
* Abutment mobility

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 7 (Estimated)
Dates: Start 2019-03-11 (Estimated); Primary Completion 2020-03-11 (Estimated); Study Completion 2020-04-11 (Estimated)

PRIMARY OUTCOMES:
Fracture | one year
  Fracture assessed by modified Ryge Criteria ( Alpha , Bravo , Charlie and Delta )

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gresnigt MM, Kalk W, Ozcan M. Clinical longevity of ceramic laminate veneers bonded to teeth with and without existing composite restorations up to 40 months. Clin Oral Investig. 2013 Apr;17(3):823-32. doi: 10.1007/s00784-012-0790-5. Epub 2012 Jul 21. PMID 22821429
- [Background] Shillingburg, H.T., Hobo, S. and Whitsett, L. (1997) Fundamentals of fixed prosthodontics. 3rd Edition, Quintessence, Chicago, 119-137, 171-174.